CLINICAL TRIAL: NCT00495053
Title: A Phase 1 Multicenter Study Evaluating the Safety and Potential Activity Of Three Escalating Doses of hMaxi-K Gene Transfer In Female Participants With Overactive Bladder Syndrome and Detrusor Overactivity: Double Blind, Imbalanced Placebo Controlled Design Within 3 Sequential Active Treatment Groups
Brief Title: Safety Study of hMaxi-K Gene Transfer to Treat Overactive Bladder and Detrusor Overactivity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment and financial issues
Sponsor: Urovant Sciences GmbH (Industry)
Collaborators: Ion Channel Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ION-02
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Overactive Bladder
Keywords: overactive bladder, urinary urgency
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: sequential, dose escalation
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- hMaxi-K 5000 µg/mL (Experimental): 5000 micrograms (µg)/90 milliliter (mL) intravesical instillation
  Interventions: Drug: hMaxi-K
- hMaxi-K 10000 µg/mL (Experimental): 10000 µg/90 mL intravesical instillation
  Interventions: Drug: hMaxi-K
- Placebo (Placebo Comparator): Matching placebo (PBS-20% sucrose)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: hMaxi-K — Two dose levels (5000 µg/90 mL intravesical instillation and 10000 µg/90 mL intravesical instillation)
  Other Names: URO-902
  Arms: hMaxi-K 10000 µg/mL; hMaxi-K 5000 µg/mL
Other: Placebo — Matching placebo (PBS-20% sucrose)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of a new product that uses human gene transfer (called hMaxi-K) when it is given to patients with overactive bladder. Human gene transfer is a new type of therapy that is the process of placing genetic material (DNA or RNA) into a person. The primary objective of this study is to evaluate safety parameters occurring subsequent to administration of a single intravesical instillation of study drug.

Two different dose groups of hMaxi-K will be tested in this study: 5000 and 10000 micrograms. A 15000 microgram group was planned; however, the study was terminated before participants were dosed. hMaxi-K will be given as a single administration into the bladder through a catheter. Each women's participation in the study will last for up to 24 weeks (followed by an additional 18-month follow-up period).

DETAILED DESCRIPTION:
The safety parameters to be monitored include: adverse events, clinical laboratory tests, electrocardiograms, and physical examinations.

The secondary objective is to evaluate the efficacy of a single intravesical instillation of hMaxi-K compared to the control group. Efficacy parameters that will be evaluated are: mean number of micturitions per 24 hours, mean number of urge incontinence episodes per 24 hours, mean number of urgency episodes per 24 hours, overall maximum bladder capacity, number of uninhibited contractions during the cystometry procedure, participant rating of urgency score, participant rating of perceived bladder condition severity, participant assessment of response to treatment, participant rating of Quality of Life (Kings Health Questionnaire), SF-12 Health Survey, International Consultation on Incontinence Questionnaire (ICIQ-SF), and pad weight measurement of accidental bladder leaks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of 18 years of age or older and of non-childbearing potential
* Clinical symptoms of overactive bladder for 6 months or longer including at least one of the following:

  1. frequent urination (that is, having to go to the bathroom 8 or more times per day);
  2. symptoms of urinary urgency, which is experiencing a sudden need to pass urine that is difficult to hold back; or the complaint of waking at night two ore more times to urinate;
  3. urge urinary incontinence, which is the complaint of leakage of urine that cannot be stopped, accompanied by or immediately preceded by urgency 5 or more times per week.
* Non-response or poor tolerance to previous treatment for symptoms of overactive bladder and do not wish to continue with that treatment.

Exclusion Criteria:

* A woman with a positive serum (HCG) pregnancy test or who is lactating
* History of three or more culture-documented recurrent urinary tract infections per year
* Current history or previous diagnosis of painful bladder syndrome (interstitial cystitis) with pain in the region of the pelvis, perineum, or lower abdomen relieved by voiding
* Current history of neurological bladder dysfunction
* A life expectancy of less than 12 months
* Current history of Grade 2 or greater cystocele
* An indwelling urethral catheter or need for clean intermittent self- catheterization
* Recent heart attack
* Uncontrolled diabetes
* Latex allergy
* Stress urinary incontinence as determined by observation of the participant coughing while standing with a full bladder and/or response of 2 or 3 on the following Stress Urinary Incontinence question: Do you experience leakage when laughing, coughing, lifting heavy objects or other types of discreet, moderately intense activities? 0=NONE: No leakage. 1=MILD: Minimal leakage on rare occasions during these types of activities; easily tolerated; do not use pads for this. 2=MODERATE: Enough leakage that it requires occasional use of pads and may interfere with usual activity and tasks. 3=SEVERE: Extreme leakage and discomfort that stops all activity and tasks and requires the use of pads on all occasions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with any treatment-emergent adverse event during the treatment period | 6 months (24 weeks per participant)
Number of participants with any treatment-emergent adverse event during the safety follow-up period | 18 months
Number of participants with any abnormal, clinically significant clinical laboratory test value during the treatment period | 6 months (24 weeks per participant)
Number of participants with any abnormal, clinically significant clinical laboratory test value during the safety follow-up period | 18 months
Number of participants with any abnormal, clinically significant clinical electrocardiogram value during the treatment period | 6 months (24 weeks per participant)
Number of participants with any abnormal, clinically significant clinical electrocardiogram value during the safety follow-up period | 18 months
Number of participants with any abnormal, clinically significant clinical physical examination finding during the treatment period | 6 months (24 weeks per participant)
Number of participants with any abnormal, clinically significant clinical physical examination finding during the safety follow-up period | 18 months

SECONDARY OUTCOMES:
Change from Baseline in the mean number of micturitions per 24 hours | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the mean number of urge incontinence episodes per 24 hours (collected over a 3-day period) | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the mean number of urgency episodes per 24 hours | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the overall maximum bladder capacity | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the number of uninhibited contractions during the cystometry procedure | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the participant rating of urgency score | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the participant rating of perceived bladder condition severity | Baseline; 6 months (24 weeks) per participant
Number of participants with the indicated response to the following question, as a measure of the participants' assessment of response to treatment: "Has the treatment been of benefit to you"? | 6 months (24 weeks) per participant
Change from Baseline in the Kings Health Questionnaire-Quality of Life (KHQ-QOL) general health perceptions domain score and impact on life domain score | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the Short Form-12 (SF-12) Health Survey | Baseline; 6 months (24 weeks) per participant
Change from Baseline in the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | Baseline; 6 months (24 weeks) per participant
Change from Baseline in pad weight | Baseline; 6 months (24 weeks) per participant

CONTACTS AND LOCATIONS:
Locations (1):
- CE3, Inc., Branford, Connecticut, United States